CLINICAL TRIAL: NCT02622893
Title: Can Surgical Approach Affect Post-operative Analgesic Requirements Following Laparoscopic Nephrectomy: Transperitoneal Versus Retroperitoneal? A Prospective Clinical Study
Brief Title: Surgical Approach Affect on Post-operative Analgesic Requirement Following Laparoscopic Nephrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Attending Anesthesiologist, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/1501
Record Dates: First submitted 2015-11-26; First posted 2015-12-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transperitoneal laparoscopic nephrectomy (Active Comparator): Patients in this group underwent transperitoneal laparoscopic nephrectomy in 45-60º modified flank position after receiving epidural catheter in the sitting position before the surgery.
  Interventions: Drug: Transperitoneal laparoscopic nephrectomy
- Retroperitoneal laparoscopic nephrectomy (Active Comparator): Patients in this group underwent retroperitoneal laparoscopic nephrectomy in lateral decubitis position after receiving epidural catheter in the sitting position before the surgery.
  Interventions: Drug: Retroperitoneal laparoscopic nephrectomy

INTERVENTIONS:
Drug: Transperitoneal laparoscopic nephrectomy — After the surgery: 10 ml 0.25% bupivacaine through epidural catheters before extubation and continuous infusion of 0,1% bupivacaine and 1 µg/ml fentanyl 5 ml/h with patient-controlled boluses of an additional 4 ml, with a lockout time of 20 min and 4-h limit of 30 ml by a patient controlled epidural analgesia (PCEA) device
  Other Names: Patient controlled epidural analgesia (PCEA)
  Arms: Transperitoneal laparoscopic nephrectomy
Drug: Retroperitoneal laparoscopic nephrectomy — After the surgery: 10 ml 0.25% bupivacaine through epidural catheters before extubation and continuous infusion of 0,1% bupivacaine and 1 µg/ml fentanyl 5 ml/h with patient-controlled boluses of an additional 4 ml, with a lockout time of 20 min and 4-h limit of 30 ml by a patient controlled epidural analgesia (PCEA) device
  Other Names: Patient controlled epidural analgesia (PCEA)
  Arms: Retroperitoneal laparoscopic nephrectomy

SUMMARY:
Background: We performed this prospective clinical study to compare the post-operative recovery profile of our patients after transperitoneal and retroperitoneal laparoscopic nephrectomy techniques. Our primary aim was to compare post-operative epidural analgesic consumption of transperitoneal (Group T) and retroperitoneal (Group R) laparoscopic nephrectomy patients within the first 24 hours.

Methods: Forty-four patients scheduled for elective transperitoneal or retroperitoneal laparoscopic nephrectomies were enrolled. All patients in both groups received epidural catheter, 2.5ml test dose of lidocaine 2% and general anesthesia induction. At the end of the surgery, patients were given 1g IV paracetamol and 10ml 0.25% bupivacaine through epidural catheters and extubated. In the post-operative care unit, patients started to receive a continuous infusion of 0,1% bupivacaine and 1µg/ml fentanyl 5ml/h with patient-controlled boluses of an additional 4ml by a patient controlled epidural analgesia (PCEA) device. They were prescribed IV tramadol 1mg/kg as a rescue analgesic (Visual analog scale (VAS)≥4). Total analgesic consumptions from PCEA devices, VAS scores at rest and during mobilization, heart rates (HRs), systolic (SBPs)/diastolic blood pressures (DBPs) at extubation (0th min-basal) and at post-operative 30th min, 2nd, 6th, 12th, 18th and 24th hours as well as number of patients who require rescue analgesic were recorded. Nausea, vomiting, time to first mobilization, return of bowel sounds and hospital stay were also documented.

DETAILED DESCRIPTION:
Background: We performed this prospective clinical study to compare the post-operative recovery profile of our patients after transperitoneal and retroperitoneal laparoscopic nephrectomy techniques. Our primary aim was to compare post-operative epidural analgesic consumption of transperitoneal (Group T) and retroperitoneal (Group R) laparoscopic nephrectomy patients within the first 24 hours.

Methods: Forty-four patients scheduled for elective transperitoneal or retroperitoneal laparoscopic nephrectomies were enrolled. All patients in both groups received epidural catheter, 2.5ml test dose of lidocaine 2% and general anesthesia induction. At the end of the surgery, patients were given 1g IV paracetamol and 10ml 0.25% bupivacaine through epidural catheters and extubated. In the post-operative care unit, patients started to receive a continuous infusion of 0,1% bupivacaine and 1µg/ml fentanyl 5ml/h with patient-controlled boluses of an additional 4ml by a patient controlled epidural analgesia (PCEA) device. They were prescribed IV tramadol 1mg/kg as a rescue analgesic (Visual analog scale (VAS)≥4). Total analgesic consumptions from PCEA devices, VAS scores at rest and during mobilization, heart rates (HRs), systolic (SBPs)/diastolic blood pressures (DBPs) at extubation (0th min-basal) and at post-operative 30th min, 2nd, 6th, 12th, 18th and 24th hours as well as number of patients who require rescue analgesic were recorded. Nausea, vomiting, time to first mobilization, return of bowel sounds and hospital stay were also documented. 0th and 30th min follow-ups were recorded in PACU and patients were passed on to ward nurses. Researchers who follow the patients at PACU and on the ward were all blinded to the surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II
* Scheduled for elective transperitoneal or retroperitoneal laparoscopic nephrectomy

Exclusion Criteria:

* Serious heart or respiratory failure
* Difficulty understanding the instructions for using the anesthetic infusion pump and/or pain scales
* Contraindications to regional anesthesia (e.g., allergy to a local anesthetics, local infection, increased intracranial pressure and coagulopathy)
* Significant neurologic disorders of the lower extremity
* Psychiatric or cognitive disorders
* History of substance abuse
* Chronic opioid use
* Patients having open nephrectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Total epidural analgesic consumption | up to 24 hours
  Total epidural analgesic (bupivacaine and fentanyl) consumption from patient controlled epidural analgesia (PCEA) devices

SECONDARY OUTCOMES:
Visual analog scale (VAS) scores | up to 24 hours
  Visual analog scale (VAS) scores at rest and during mobilization
Number of patients who require rescue analgesic | up to 24 hours
  Number of patients who require IV tramadol (1 mg/kg) as a rescue analgesic besides PCEA use
Hemodynamic parameters | up to 24 hours
  Postoperative heart rates (HRs), systolic (SBPs)/diastolic blood pressures (DBPs)

OTHER OUTCOMES:
Complications | up to 24 hours
  Nausea, vomiting
Time to first mobilization | up to 24 hours
  Time to first mobilization
Return of bowel sounds/oral intake | through study completion, an average of 1 week
  Post-operative oral intake starts just after the return of bowel sounds (almost at the same time), will be assessed as hours (time to return of bowel sounds)
Hospital stay | through study completion, an average of 1 week
  Hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Department of Anesthesiology, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Savran-Karadeniz M, Kisa I, Salviz EA, Ozkan-Seyhan T, Tefik T, Sanli O, Tugrul KM. Can surgical approach affect postoperative analgesic requirements following laparoscopic nephrectomy: Transperitoneal versus retroperitoneal? A prospective clinical study. Arch Esp Urol. 2017 Jul;70(6):603-611. PMID 28678012